CLINICAL TRIAL: NCT02611063
Title: A Phase I Trial of Fostamatinib and Chronic Graft vs. Host Disease Development After Allogeneic Stem Cell Transplantation
Brief Title: Evaluation of Fostamatinib in Patients With cGVHD After Allogeneic Stem Cell Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stefanie Sarantopoulos, MD, PhD. (Other)
Responsible Party: Sponsor-Investigator, Stefanie Sarantopoulos, MD, PhD., Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00064227
Record Dates: First submitted 2015-11-16; First posted 2015-11-20 (Estimated); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Hematological Malignancies
Keywords: allogeneic stem cell transplant
MeSH Terms: conditions — Hematologic Neoplasms | interventions — fostamatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fostamatinib (Experimental): Subjects will receive fostamatinib 100 mg qd, 150 mg qd, or 100 mg bid with dosage determined by the modified continual reassessment method. The treatment period begins at baseline 90 days after transplant and continues for up to 1 year after transplant. In patients with steroid-refractory cGVHD who are also included on this study, these subjects also receive fostamatinib 100mg qd, 150mg qd, or 100mg bid dosage determined by the modified continual reassessment method.
  Interventions: Drug: fostamatinib

INTERVENTIONS:
Drug: fostamatinib — 100mg qd, 150mg qd, or 100mg bid

SUMMARY:
The purpose of this study is to evaluate whether fostamatinib, a drug that blocks activated B cells will be effective in preventing and treating chronic graft vs host disease (cGVHD) after allogeneic stem cell transplant. Activated B cells may play a role in development of cGVHD. Inhibiting the B cell activation using fostamatinib after allogeneic stem cell transplant may prevent the development of cGVHD.

DETAILED DESCRIPTION:
Design & Procedures

All patients will undergo allogeneic stem cell transplantation (HCT) according to the program's standards. No specific conditioning regimen is mandated. The stem cell source must have been peripheral blood stem cells. Prophylaxis against acute GVHD must be with standard agents (sirolimus and/or tacrolimus and/or methotrexate and/or cyclosporine). Participation in a trial evaluating novel agents for therapy of acute GVHD is allowed, as long as the experimental agent was discontinued > 14 days prior to trial entry.

Therapy: Patients will receive 100mg daily, 150mg daily or 100 mg bid beginning 90 days after allogeneic transplantation and continue for up to 1 year from day of transplant OR beginning at time of steroid-refractory cGVHD. Dosage will be determined using the modified continual reassessment method.

Patient evaluations: Patients will be evaluated for cGVHD and other toxicity at a minimum on day 1(baseline), day 3, day 11, day 25, day 39, day 60, day 88, day 116, day 144, day 186, day 228, and day 275 from initiation of protocol therapy. While the assessment for safety is determined based on the evaluation at day 60, patients may stay on therapy for up to 1 year after transplantation (study treatment day 275). In addition, patients will be observed for one year after stopping study treatment with evaluation for toxicity and cGVHD during clinic visits at 6 and 12 months after completion of study therapy. If at any time within the first year after transplantation, a study subject is determined to have evidence of moderate or severe stage cGVHD according to NIH consensus criteria for global severity, the subject will be removed from this clinical trial and appropriate therapy for cGVHD will be administered per the treating physician's discretion. The study subject may continue to receive Fostamatinib as per the guidelines of this clinical trial in the event that mild stage cGVHD is diagnosed. If cGVHD develops during the observation period, a second course of Fostamatinib at 100% tolerated study dose may be given during the observation period.

Immunosuppressive and other medications should be tapered according to the treating physicians' discretion with careful attention to the clinical trial or treatment plan to which the participating subject is already enrolled.

Laboratory samples will be obtained according to the study schedule. The following tests are to be collected and analyzed for the study: complete blood counts, serum chemistry, liver function tests (LFTs), chimerism analysis if indicated, and immunology/correlative science studies.

This study will be open to members of all demographic groups who meet the eligibility criteria. Approximately 18 subjects will be recruited at Duke.

A total of eighteen patients will receive fostamatinib beginning at day 90 after allogeneic transplantation. The safety assessment is determined at day 60. Patients with steroid-refractory cGVHD are also eligible for this phase I study. Three dose levels are considered: 100 mg qd, 150 mg qd, 100 mg bid, and the target dose-limiting toxicity (DLT) probability is 0.33. The Bayesian model averaging continual reassessment method (BMA-CRM) will be used for this trial.[15]

The investigators will study targeted molecular mechanisms underpinning aberrant B-cell signaling in cGVHD. Corollary studies will determine whether B and T cell subsets and/or soluble B-cell activation factors are altered after Syk inhibition. The objective is to implement preemptive targeted therapies that decrease excessive immune activation in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have undergone allogeneic stem cell transplantation for the treatment of any hematological malignancy are eligible. Transplant must have occurred 90 days before the start of study drug.
2. Peripheral blood stem cells must have been used as the stem cell source.
3. Patients must have received transplantation from adult donors (both related and unrelated) who are Human Leukocyte Antigen (HLA) matched or mismatched at 1 locus (5/6) or are mismatched at one allele (3/6). Class I and II typing is to be performed by standard methods at our institution.
4. Complete remission of hematological malignancy prior to transplantation. All patients must have undergone appropriate staging for their malignancy prior to transplantation including bone marrow aspirate/biopsy and radiographic scanning if indicated.
5. Patients who have undergone a non-myeloablative stem cell transplant must have > 65% donor lymphoid hematopoiesis within 30 days of study enrollment.
6. Patient age greater than 18 years of age.
7. ECOG performance status 0-2 or Karnofsky Performance Status (KPS) > 60.
8. Must be able to tolerate routine oral posaconazole or voriconazole as fungal prophylaxis therapy.
9. Written informed consent.

Exclusion Criteria:

1. Recipients of allogeneic stem cell transplantation using a single or multiple umbilical cord blood units or using bone marrow.
2. Participation in a clinical trial evaluating another preventative strategy for chronic GVHD or ongoing participation in a clinical trial for therapy of acute GVHD. Prior completion of experimental therapy for acute GVHD is permissible if the experimental agent was used > 14 days prior to enrollment.
3. Evidence of relapsed hematologic malignancy based on routine restaging studies.
4. Evidence of any active uncontrolled infection (bacterial, viral or fungal) or evidence of natural exposure to Hepatitis B, Hepatitis C or HIV without demonstration of PCR negativity for said virus. Vaccination to Hepatitis B is not an exclusion criterion.
5. Any evidence of ongoing gastrointestinal or hepatic acute GVHD or evidence of greater than ongoing Stage I cutaneous acute GVHD at time of enrollment. Ongoing, tapering therapy for resolved acute GVHD is permissible.
6. Patients with GVHD with chronic features diagnosed prior to day +60 or prior to enrollment are ineligible.
7. Patients may have received no more than one Donor Lymphocyte Infusion (DLI), DLI must have been administered > 6 weeks prior to enrollment on study, and no plans for a DLI in the upcoming 30 days.
8. Any major cardiovascular even within 6 months of study initiation, including but not limited to myocardial infarction, unstable angina, cerebrovascular accident, pulmonary embolism, heart failure uncontrolled by medications or New York Heart Association Class III or IV heart failure.
9. Uncontrolled or poorly controlled hypertension, defined as systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg, whether or not the subject is receiving anti-hypertensive treatment. Subjects may be rescreened if the blood pressure is successfully and promptly controlled within 5 days using conventional anti-hypertensive therapy to achieve optimal blood pressure control (<140/90 mmHg).
10. Active hemolytic anemia.
11. History of arterial or venous thrombosis (unless a single episode of venous thrombosis > 1 year prior to study initiation).
12. Liver function test abnormalities including ALT or AST > 3.0x ULN; total bilirubin > 1.5x ULN; alkaline phosphatase > 2.5 x ULN
13. Neutrophil count < 1.5 x 10e9/L or platelet count < 75 x10e9/L
14. Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-01; Primary Completion 2021-02 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Evaluate maximum tolerated dose of fostamatinib delivered following allogenic transplantation | day 60 after fostamatinib initiation
  three dose levels are considered: 100 mg qd, 150 mg qd, 100 mg bid dose limiting toxicity is any of the following
  1. Grade > or = II aGVHD of the gut or liver or Grade III aGVHD of the skin lasting > 7 days and related to the agent
  2. Grade 3 toxicity from the agent in the cardiac, dermatologic, gastrointestinal, hepatic, pulmonary, renal/genitourinary or neurologic categories that lasts > 5 days
  3. fostamatinib related mortality (TRM)
  4. absolute neutrophil count (ANC) of Grade 3 or 4 plus fever attributable to the agent
  5. ANC<0.5 x 10e9/L for >5 days and attributable to the agent
  6. platelet < 25 x 10e 9/L and attributable to the agent

SECONDARY OUTCOMES:
Incidence of chronic graft vs host disease (cGVHD) | one and two years when fostamatinib administered after allogeneic HCT
Incidence of relapse of chronic graft vs host disease (cGVHD) | one and two years when fostamatinib administered after allogeneic HCT
B-cell activation rate | two years
  B-cell activation rate before and after fostamatinib administration
B-cell death rate | two years
  B-cell death rate before and after fostamatinib administration
Number of B-cells | two years
  Immune recovery as measured by the number of B-cells before and after fostamatinib administration

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Sarantopoulos, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University of Medicine, Durham, North Carolina, United States